CLINICAL TRIAL: NCT06245993
Title: Study of Residuals Deformities After Diaphyseal Femoral Fracture in Children Treated by Skin Traction
Acronym: FRAFEMKID
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0060
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: EOS
Keywords: EOS; skin traction; femoral fracture; remodeling; leg length
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diaphyseal femoral fracture treated children
  Interventions: Other: EOS imaging

INTERVENTIONS:
Other: EOS imaging — EOS imaging 3 years after skin traction treatment for femoral shaft fracture.

SUMMARY:
Diaphyseal femoral fracture in children <6 years old are treated by the skin traction technique. As demonstrated by numerous studies, given the significant potential for bone remodeling in young children, remodeling (excluding rotational disorder) allows anatomical correction. The aim of this study is to confirm, via EOS imaging, the absence of residual deformities 3 years after the end of treatment in children treated in Amiens hospital department.

ELIGIBILITY:
Inclusion Criteria:

* <6 years old at the time of the fracture
* treatment by skin zenith traction
* femoral shaft fracture, traumatic, unilateral

Exclusion Criteria:

* Multiple fracture
* pathological fracture
* history of lower limb fracture
* contraindication to zenith traction

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diaphyseal femoral fracture in children <6 years old are treated by the skin traction.
  The children have a Clinical examination and EOS imaging 3 years after skin traction treatment for femoral shaft fracture.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
absence of lower limb overgrowth | 3 years
  Leg Length Discrepancy in EOS imaging

SECONDARY OUTCOMES:
Measurement of the angle on the lower limb sagittal axis | 3 years
  Measurement of the angle on the sagittal axis of the lower limb 3 years after the end of treatment
Measurement of the angle on the lower limb on the frontal axis | 3 years
  Measurement of the angle on the frontal axis of the lower limb 3 years after the end of treatment
Measurement of the angle on the lower limb on the frontal axis | 3 years
  Measurement of the angle on the femoral torsion of the lower limb 3 years after the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No